CLINICAL TRIAL: NCT02556645
Title: A Comparison of Web-Prolonged Exposure (Web-PE) and Present-Centered Therapy (PCT) for PTSD Among Active-Duty Military Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Texas (Other); VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Carmen McLean, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-14-1-0008; 12012005 (Other: Department of Defense)
Record Dates: First submitted 2015-07-24; First posted 2015-09-22 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Posttraumatic Stress Disorders; Combat Disorders
Keywords: Combat; Psychological Treatment; Military; Psychotherapy; Trauma; Posttraumatic Stress; Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Web-PE (Experimental): Ten 60-minute psychotherapy sessions over 8 weeks, focused on gradually confronting distressing trauma-related memories and reminders. Web-PE is an internet-based version of prolonged exposure (PE) for posttraumatic stress disorder (PTSD).
  Interventions: Other: Web-PE Therapy
- PCT (Active Comparator): Ten 60-minute psychotherapy sessions over 8 weeks, focused on identifying and solving day-to-day problems as they are brought up by the participants. PCT is a manualized therapy that has been used as active control condition in several CBT studies.
  Interventions: Other: Therapist-Delivered Present-Centered Therapy

INTERVENTIONS:
Other: Web-PE Therapy — Ten 60-minute psychotherapy sessions over 8 weeks, focused on gradually confronting distressing trauma-related memories and reminders. Web-PE is an internet-based version of prolonged exposure (PE) for posttraumatic stress disorder (PTSD).
  Other Names: Internet-based prolonged exposure
  Arms: Web-PE
Other: Therapist-Delivered Present-Centered Therapy — Ten 60-minute psychotherapy sessions over 8 weeks, focused on identifying and solving day-to-day problems as they are brought up by the participants. PCT is a manualized therapy that has been used as active control condition in several CBT studies. It provides a credible comparison therapy to control for nonspecific therapeutic factors so that observed effects of Web-PE can be attributed to its specific ingredients beyond the benefits of good therapy.
  Other Names: PCT
  Arms: PCT

SUMMARY:
The purpose of this randomized controlled trial is to compare the efficacy and potential biological mechanisms of action of 10 sessions of a web-version of Prolonged Exposure (PE), "Web-PE," delivered over 8-weeks to 10 sessions of Present Centered Treatment (PCT) delivered over 8-weeks by a therapist in 120 active duty military personnel with PTSD. Up to 170 individuals will be consented to obtain data from 120 for analysis. Participants will be assessed at pre-treatment, mid-treatment, and 1-, 3- and 6-months after treatment completion.

DETAILED DESCRIPTION:
Background: It is urgent to make EBTs for military personnel readily accessible in order to meet the growing demand for effective and efficient treatment for PTSD in a timely manner. Effective EBTs for PTSD are available, but barriers to accessing care can deter military personnel from accessing care. Web-treatments represent an innovative way to overcome these barriers. The efficacy of previously developed web-treatments for PTSD appear promising, however, they are not based on treatment protocols with strong empirical support for their efficacy. Hence, it cannot be discerned whether the outcomes associated with existing web-treatments are due to the new intervention or to factors associated with the use of the Internet to deliver the treatment. No study to date has examined web-treatment of PTSD using a well-established treatment program. An important unanswered question is whether moving from the traditional, costly, access-limiting, therapist-delivered format of an effective treatment to a more accessible, cost-effective, web-format will impact treatment efficacy. In addition, based on evidence showing a link between neurosteroids and psychopathology and a role in PTSD treatment response, an add-on biomarkers study was funded that examines the role of candidate biomarkers [endogenous glucocorticoids and neurosteroids, i.e. cortisol, allopregnanolone (ALLO) and metabolites, and dehydroepiandrosterone (DHEA/DHEAS)] as: a) predictors of treatment response, and b) indices of therapeutic change during PTSD treatment.

Objective/Hypotheses: To eliminate the confound inherent in changing simultaneously both the treatment program and the mode of delivery, the investigators propose to develop a web-version of PE, "Web-PE", and compare its efficacy to Present Centered Treatment (PCT), an active control comparison. The investigators hypothesize that Web-PE will be a more efficacious in reducing PTSD severity than PCT among military personnel returned from deployments in Afghanistan and Iraq at post-treatment and 3- and 6-months after treatment completion. In addition, the investigators expect that changes cortisol and neurosteriods will track symptom change.

Specific Aims: The first aim is to develop a Web-PE program that will receive high ratings of ease of use, acceptability, comprehension of program content and functionality, and overall satisfaction by military personnel with PTSD symptoms and an advisory board of eight experts in PE and the treatment PTSD in the military. The second aim is to examine the efficacy of Web-PE by comparing it to therapist-delivered PCT on the following outcomes: 1) Change in PTSD severity and diagnostic status from pre- to post-treatment; 2) Change in symptoms of depression, anger, and other frequently co-occurring problems from pre- to post-treatment. The biological aims of the study include: 1) To identify specific neuroendocrine and neurosteroid changes that "track" Posttraumatic Stress Disorder (PTSD) symptom change over the course of effective treatment and 2) to determine the specificity of Prolonged Exposure (PE) -induced neuroendocrine/neurosteroid changes by directly comparing patterns of change during PE to those during Present Centered Therapy (PCT).

Study Design: During Phase I (months 0-9), the investigators will develop and demonstrate the feasibility of the Web-PE program by piloting it with 10 military personnel with PTSD or subclinical PTSD and by members of the expert advisory board. During Phase II (months 9-36), the investigators will conduct an RCT comparing the efficacy of Web-PE with therapist-delivered PCT on measures of PTSD symptom severity and related psychopathology with 160 OIF/OEF active duty military personnel with PTSD. Cortisol Awakening Response collected at home on the three mornings prior to the research sessions that occur at baseline, week 4, one and three months follow-up. Script driven imagery saliva collection for salivary cortisol in response to the general environment and specific trauma cues at baseline, week 4, and one and three months follow-up. Serum neurosteriods (allopregnanolone, pregnenolone, pregnanolone, androsterone, DHEA) at baseline, week 4 and 1 month follow-up of treatment.

Relevance: Untreated PTSD becomes a chronic disorder, leaving military service-men and -women less effective or unable to perform their military duties, more likely to have comorbid mental and physical health problems as well as difficulties in daily functioning (Vasterling et al., 2007). The proposed Web-PE program can function as the first step in a step care model. As such it is expected to greatly facilitate the dissemination of EBT to those in need by capitalizing on the greater accessibility, cost-effectiveness, and anonymity that is afforded by Internet. Thus, the proposed study directly targets the MOM/JPC interest in research aim at developing and validating novel EBTs that exploit innovative telemedicine technologies. Because Web-PE could be accessed at home, the proposed study is also relevant to the MOM/ JPC interest in strategies to reduce the stigma associated with PTSD treatment. Integrating affective neuroscience methods into an RCT can make each study more informative, effective, and less expensive than two independent studies. Neurobiological studies of PTSD have linked specific candidate biomarkers [endogenous glucocorticoids and neurosteroids, i.e. cortisol, allopregnanolone (ALLO) and metabolites, and dehydroepiandrosterone (DHEA/DHEAS)] to PTSD severity and potentially to treatment response. Identifying the mechanisms involved in treatment response can assist in improving therapeutic techniques by targeting specific neurobiological processes involved.

This study is affiliated with the South Texas Research Organizational Network Guiding Studies on Trauma and Resilience (STRONG STAR) (Consortium Director: Alan L. Peterson, Ph.D., ABPP, Professor, Behavioral Wellness Center for Clinical Trials, Department of Psychiatry-Mail Code 7792, University of Texas Health Science Center at San Antonio (UTHSCSA), 7703 Floyd Curl Drive, San Antonio, TX 78229-3900). The Overall PIs for this study are Carmen P. McLean, Ph.D. of the Center for the Treatment and Study of Anxiety at the University of Pennsylvania and, for the biological measures portion of the study, Sheila Rauch, Ph.D., ABPP of Emory University. The PI for this study at the University of Texas Health Science Center at San Antonio (UTHSCSA) is Alan Peterson, Ph.D., ABPP, Department of Psychiatry, Division of Behavioral Medicine. The on-site PI is COL Jeffrey Yarvis, Ph.D.,Chief, Soldier Behavioral Health/Outpatient Psychiatry, Carl R. Darnall Army Medical Center, 36000 Darnall Loop, Fort Hood, TX, 76544. The study will be conducted at Fort Hood, Texas.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female active duty military personnel or veterans who have deployment since 9/11, ages 18-65 seeking treatment for PTSD. Veterans must be eligible for military medical care on Fort Hood.
* Diagnosis of PTSD as determined by a Clinician Administered PTSD Scale for DSM-5 (CAPS-5) clinical interview score ≥ 25. Person has experienced a Criterion A event that is a specific combat-related event or high magnitude operational experience that occurred during a period of recent military deployment. The diagnosis of PTSD may be indexed to that event or to another Criterion A event.
* Able to speak and read English
* Indication that the participant plans to be in the area for the next five months following the first assessment

Exclusion Criteria:

* Recent manic episode (past 12 months) or a psychotic disorder (as determined by the bipolar and psychosis sections of the MINI)
* Current alcohol dependence (as determined by an a score of ≥ 4 on items #4-6 and a total score of ≥20 on the AUDIT)
* Evidence of a moderate or severe traumatic brain injury (as determined by the inability to comprehend the baseline screening questionnaires)
* Current suicidal ideation severe enough to warrant immediate attention (as determined by the Depressive Symptoms Index-Suicidality Subscale and corroborated by a clinical risk assessment by a credentialed provider)
* Other psychiatric disorders severe enough to warrant designation as the primary disorder
* Recent course of PE within the past 12 months
* Currently engaged in evidence-based treatment for PTSD (e.g. Prolonged Exposure Therapy or Cognitive Processing Therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05; Primary Completion 2018-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of Web-PE relative to PCT in the reduction of PTSD severity (using the CAPS severity score). | Three years
To evaluate the efficacy of Web-PE relative to PCT in the reduction in associated psychopathology | Three years
  Associated psychopathology: PTSD diagnosis and severity scores on measures of depression, general anxiety, anger, and PTSD-related cognitions
To evaluate the efficacy of Web-PE relative to PCT in the change in associated biomarkers | Three years
  i.e., Cortisol response to awakening, cortisol response to script-driven imagery, salivary and serum neurosteroids.

SECONDARY OUTCOMES:
Composite ratings on the use of the Web-PE program | Three years
  Ratings of ease of use, acceptability, comprehension of program content and functionality, and overall satisfaction of the Web-PE program. Ratings made by military personnel with PTSD symptoms and an advisory board of eight experts in PE and the treatment PTSD in the military.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen McLean, Ph.D., Principal Investigator — University of Pennsylvania; Sheila Rauch, Ph.D., Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Department of Psychiatry and Behavioral Sciences, Emory University, Atlanta, Georgia
  - Center for the Treatment and Study of Anxiety, University of Pennsylvania, Philadelphia, Pennsylvania
  - Carl R. Darnall Army Medical Center, Killeen, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- See also: Link to STRONG STAR research consortium — https://tango.uthscsa.edu/strongstar/